CLINICAL TRIAL: NCT01838525
Title: Alpha-1-acid Glycoprotein as a Biomarker of Developmental Diagnosing and Monitoring Effectiveness in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Longxiang Su, Attending Doctor, Chinese PLA General Hospital
Other Study IDs: 20130419-007
Record Dates: First submitted 2013-04-19; First posted 2013-04-24 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Systemic Inflammatory Response Syndrome; Sepsis
Keywords: sepsis; alpha-1-acid glycoprotein (AGP); diagnosis; prognosis; SIRS
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Sepsis; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- SIRS, SEPSIS
- sepsis, severe sepsis, septic shock
- health, SIRS, Sepsis

SUMMARY:
To assess the potential value of alpha-1-acid glycoprotein (AGP) for early diagnosis and prognosis of patients with sepsis, and then compared with C-reactive protein (CRP), procalcitonin (PCT), white blood cell (WBC) counts, Acute Physiology and Chronic Health Evaluation (APACHE) II score and Sequential Organ Failure Assessment (SOFA) score. 164 patients were enrolled in the study, including 25 cases with systemic inflammatory response syndrome (SIRS) and 139 cases with different levels of sepsis (46 moderate sepsis, 52 severe sepsis and 41 septic shock ). Serum levels of Alpha-1-acid Glycoprotein (AGP), C-reactive protein (CRP), and procalcitonin (PCT), and white blood cell (WBC) counts were measured on the day of admission to intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18 years old and over;
2. Clinically suspected infection;
3. Fulfilled at least two criteria of systemic inflammatory response syndrome (a) core temperature higher than 38 °C or lower than 36 °C (b)respiratory rate above 20/min, or PCO2 below 32 mmHg (c) pulse rate above 90/min, and (d) white blood cell count greater than 12,000/μl or lower than < 4,000/μl or less than 10% of bands;

Exclusion Criteria:

1. less than 18 years old;
2. immunosuppression;
3. agranulocytosis (granulocyte counts <0.5× 109/L);
4. chronic myeloid leukemia (CML);
5. malignancy;
6. less than 24 hours of the length of ICU stay;
7. reluctant to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between April 2011 and APRIL 2013, inpatients were included who were in the intensive care units (ICU) of the Department of Respiratory Disease (RICU), the Emergency Department (EICU), and the Department of Surgery (SICU) of the Chinese People's Liberation Army General Hospital.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2011-04; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Patients Outcome | 28 days
  The survival time of patients more than 28 days is defined as survival. The survival time of patients less than 28 days is defined as death

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, doctor, Study Director — Department Of Respiratory Diseases, Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Xiao K, Su L, Yan P, Han B, Li J, Wang H, Jia Y, Li X, Xie L. alpha-1-Acid glycoprotein as a biomarker for the early diagnosis and monitoring the prognosis of sepsis. J Crit Care. 2015 Aug;30(4):744-51. doi: 10.1016/j.jcrc.2015.04.007. Epub 2015 Apr 17. PMID 25957497